CLINICAL TRIAL: NCT05158725
Title: Comparison of Colonoscopy Adenoma Detection Yield of Standard Colonoscopy, Discovery Aided Colonoscopy, and Discovery and G-EYE® Aided Colonoscopy
Brief Title: Comparison of Colonoscopy Adenoma Detection Yield
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Horst Schmidt Klinik GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: G-EYE/Discovery
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Adenoma Colon

STUDY DESIGN:
Intervention Model Description: Multi-center, three-arm, randomized, controlled, open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Colonoscopy (Active Comparator): Subjects will undergo colonoscopy using a standard colonoscope
  Interventions: Device: Standard Colonoscopy
- Discovery aided colonoscopy (Active Comparator): Subjects will undergo colonoscopy using a a standard colonoscope and the Discovery aided colonoscopy
  Interventions: Device: Discovery aided colonoscopy
- Discovery and G-EYE aided colonoscopy (Experimental): Subjects will undergo colonoscopy using the G-EYE Endoscope and the Discovery aided colonoscopy
  Interventions: Device: Discovery and G-EYE

INTERVENTIONS:
Device: Standard Colonoscopy — In this arm, subjects will undergo colonoscopy using a standard colonoscope
  Arms: Standard Colonoscopy
Device: Discovery aided colonoscopy — the Discovery is a customized detection support software, developed utilizing AI deep learning technology to support endoscopic lesion detection in the colon. In this arm, a standard colonoscope is used with the Discovery.
  Arms: Discovery aided colonoscopy
Device: Discovery and G-EYE — The G-EYE® Endoscope is a standard colonoscope which is remanufactured by installing the G-EYE® balloon on the distal bending section of the colonoscope. in this arm, the G-EYE® Endoscope is used with the Discovery
  Arms: Discovery and G-EYE aided colonoscopy

SUMMARY:
A Prospective Randomized Comparison of colonoscopy Adenoma Detection Yield of (i) Standard Colonoscopy (SC), (ii) artificial intelligence (Discovery) aided colonoscopy, and (iii) artificial intelligence (Discovery) and permanently mounted balloon (G-EYE®) aided colonoscopy.

DETAILED DESCRIPTION:
Multi-center, three-arm, randomized, controlled, open-label study.

Total of up to 1320 patients will be randomized, including up to 10% for subject drop-out, 440 to each of the three following arms (groups):

Group 1 (1st arm): patients will receive standard colonoscopy (SC) Group 2 (2nd arm): patients will receive colonoscopy aided by the Discovery artificial intelligence software (DC) Group 3 (3rd arm): patients will receive colonoscopy aided by the Discovery artificial intelligence software and the G-EYE® balloon (GDC) The purpose of this study is to compare between the diagnostic yield of Standard Colonoscopy, Discovery aided colonoscopy, and Discovery & G-EYE® aided colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Screening and surveillance population for Adenoma and CRC.
2. The patient must understand and sign a written informed consent for the procedure.

Exclusion Criteria:

1. Subjects with inflammatory bowel disease;
2. Subjects with a personal history of hereditary polyposis syndrome;
3. Subjects with suspected chronic stricture potentially precluding complete colonoscopy;
4. Subjects with diverticulitis or toxic megacolon;
5. Subjects with prior colonic surgery (exclusion appendectomy)
6. Subjects with a history of radiation therapy to abdomen or pelvis;
7. Pregnant or lactating female subjects;
8. Subjects who are currently enrolled in another clinical investigation.
9. Subjects with current oral or parenteral use of anticoagulants, not considered eligible by the investigator.
10. Subjects with recent (within the last 3 mounts) coronary ischemia or CVA (stroke)
11. Any patient condition deemed too risky for the study by the investigator

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1320 (Estimated)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection yield | Upon histology results (up to 30 days)
  adenoma detection yield, represented by Adenoma Per Colonoscopy (APC), of Standard Colonoscopy, compared with APC of Discovery aided colonoscopy and further compared with APC of Discovery & G-EYE® aided colonoscopy

SECONDARY OUTCOMES:
Adenoma Detection Rate (Discovery + G-EYE vs. Standard Colonoscopy) | Upon histology results (up to 30 days)
  Adenoma Detection Rate of Discovery and G-EYE® aided colonoscopy compared to Adenoma Detection Rate of Standard Colonoscopy
Adenoma Detection Rate (Discovery vs. Standard Colonosocopy) | Upon histology results (up to 30 days)
  Adenoma Detection Rate of Discovery aided colonoscopy compared to Adenoma Detection Rate of Standard Colonoscopy
Adenoma Per Colonoscopy (Discovery vs. Discovery + G-EYE) | Upon histology results (up to 30 days)
  Adenoma Per Colonoscopy of Discovery aided colonoscopy compared to Adenoma Per Colonoscopy of Discovery and G-EYE® aided colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Kiesslich, Prof., Principal Investigator — Helios Dr. Horst Schmidt Kliniken Wiesbaden GmbH
Locations (1):
- Helios Dr. Horst Schmidt Kliniken Wiesbaden GmbH, Wiesbaden, Germany

IPD SHARING:
Plan to Share IPD: Undecided